CLINICAL TRIAL: NCT06114030
Title: Clinical and Radiographical Evaluation of CAD-CAM Crowns With and Without Deep Margin Elevation: Up to 10-year Results
Brief Title: Clinical and Radiographical Evaluation of CAD-CAM Crowns With and Without Deep Margin Elevation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ahmed Aziz, Assistant Professor, University of Sharjah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50571100
Record Dates: First submitted 2023-10-17; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Caries,Dental; Crown of Tooth With Poor Contour; Broken Teeth; Survival, Prosthesis; Failure, Prosthesis
MeSH Terms: conditions — Dental Caries; Tooth Fractures; Prosthesis Failure | interventions — Composite Resins; Tetric EvoCeram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep margin elevation followed by crowns (Other): Teeth restored with DME and crowns
  Interventions: Procedure: Deep margin elevation with composite resin and Lithium disilicate glass-ceramic crowns

INTERVENTIONS:
Procedure: Deep margin elevation with composite resin and Lithium disilicate glass-ceramic crowns — Restoration of the deep margin by composite restorations such as: Filtek Supreme XTE, Tetric EvoCeram, Estelite Sigma Qquick followed by Lithium disilicate glass-ceramic CAD/CAM crowns (IPS e.max CAD).
  Other Names: Filtek Supreme XTE (3M ESPE, Seefeld, Germany); Tetric EvoCeram (Ivoclar Vivadent AG, Schaan, Lichtenstein); Estelite Sigma Qquick (Tokuyama, Tokyo, Japan); IPS e.max CAD (Ivoclar Vivadent AG, Schaan, Lichtenstein)

SUMMARY:
Deep margin elevation (DME) is a non-invasive restorative technique to relocate the deep cervical margin to a supragingival position using resin composite. This retrospective multicenter practice-based study will assess the long-term clinical performance and periodontal health of teeth restored with CAD-CAM crowns with or without DME. Patients who will receive CAD-CAM lithium disilicate (LD) crowns with or without DME between 2013 and 2023 at multiple private practices will be included. When indicated, DME will be performed using resin-based restoration. Clinical assessment of the crowns and supporting periodontal structures will be performed following the modified United States Public Health Service (USPHS) criteria. Intra-oral photographs, periapical and bitewing radiographs will be taken for further assessment by three evaluators. Kaplan Meier survival analyses will be performed.

DETAILED DESCRIPTION:
The ethical approval to conduct this retrospective multicenter practice-based study was obtained from the Research Ethics Committee at the University of Sharjah (REC-23-09-11-01-F). The present report will complie with the STROBE guidelines for cohort studies.

Participants selection Patient records at 7 private practices in the UAE will be searched for the presence of posterior LD CAD-CAM crowns during 2013 to 2016. Inclusion criteria: adult patient and indication for crown with or without DME. Exclusion criteria: poor oral hygiene and active periodontal disease. A total of 560 eligible patients will be invited to a clinical examination.

Clinical Examination The clinical evaluation will be conducted by three calibrated independent prosthodontists. Patients will be requested to read and sign an informed consent form to participate in the study. Intraoral photographs, Periapical and bitewing radiographs will be obtained to assess the emergence profile of the DEM which should ideally reproduce the normal morphology. Both the crowned tooth and the contralateral tooth were assessed clinically for the following parameters: pocket depth (PD), BoP, and presence of plaque using a plaque indicator liquid (Mira-2 Ton Liquid, Hager & Werken; Duisburg, Germany). Bone level will be assessed by comparing a measurement from the margin of the tooth to the crest of the bone on bitewing radiographs to corresponding preoperative radiographs.

A comprehensive assessment of the restored teeth will be carried out following the modified United States Public Health Service (USPHS) criteria. The location of crown margin will be recorded clinically and radiographically to assess the association between periodontal health and margin location. The primary outcomes will be the survival rate and time to event. The secondary outcome will be the success rate. The success is defined as a crown that had remained unchanged over the observation period, while survival is defined as a crown that was in situ at the examination visit but might exhibits chipping or have been repaired. Failure will be scored for the followings: recurrent caries, loss of vitality, tooth fracture, and crown fracture.

Statistical analysis Descriptive statistics were computed with a statistical software program (IBM SPSS Statistics, v29; IBM Corp., Armonk, NY, USA). Each complication will be considered as a statistical event. The statistical testing will be 2-tailed (a=.05). The McNemar chi-squared and Fisher exact tests will be used to assess the severity of PD, BoP and plaque deposition. Odds ratios and their 95% confidence intervals will be reported. The Pearson chi-squared test for differences in proportions will be used to assess the relationship between the location of margins and the associated condition of the periodontal tissues. Kaplan-Meier survival analysis will be performed to calculate the overall crown survival and success probabilities. Cox regression models will be used to evaluate the effect of various confounding factors on the survival and success rates.

ELIGIBILITY:
Inclusion Criteria: :

* adult patient and indication for crown with or without DME.

Exclusion Criteria:

* poor oral hygiene and active periodontal disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The survival rate of teeth restored with or without DME and crowns. | 10 years
  Number of survived crowns in the presence or absence of DME
Number of failed crowns in the presence or absence of DME | 10 years

SECONDARY OUTCOMES:
Change from baseline in pocket depth | 10 years
Change from baseline in bleeding of probing | 10 years
Periodontal responses in response to deep (subgingival) margins | 10 years
  Change from baseline in bone level cervically

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Aziz, PhD, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No